CLINICAL TRIAL: NCT07043153
Title: Using Combination of Albumin to Globulin Ratio and Prognostic Nutritional Index Model for Predicting Disease Activity in Patients With Systemic Lupus Erythematosus
Brief Title: AGR+PNI as Predictors of Systemic Lupus Erythematosus Disease Activity
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hala Abdellatif Hamed, Resident of Physical Medicine, Rheumatology and Rehabilitation Department, Sohag University
Other Study IDs: Soh-Med--25-6-1MS
Record Dates: First submitted 2025-06-19; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Systemic Lupus Erythematosus Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active SLE group:patients with active (SLE), fulfilling the ACR/EULAR classification criteria,
  Interventions: Diagnostic Test: Albumin to globulin ratio and prognostic nutritional index model
- Healthy controls:Age and sex-matched healthy individuals without any history of autoimmune diseases
  Interventions: Diagnostic Test: Albumin to globulin ratio and prognostic nutritional index model

INTERVENTIONS:
Diagnostic Test: Albumin to globulin ratio and prognostic nutritional index model — Measurement of albumin to globulin ratio and prognostic nutritional index in participants to assess disease activity in systemic lupus erythematosus patients

SUMMARY:
This study aims to evaluate the clinical utility of combining the albumin to globulin ratio (AGR) and the prognostic nutritional index (PNI) as a predictive model for assessing disease activity in patients with systemic lupus erythematosus (SLE). By correlating these nutritional and inflammatory markers with clinical manifestations and laboratory parameters, we hope to establish a simple, non-invasive, and cost-effective tool to aid in monitoring disease activity in Systemic lupus erythematosus patients.

ELIGIBILITY:
Inclusion Criteria:

* · Age ≥ 18 years.

  * Both sexes.
  * Patients diagnosed with SLE who fulfilling the Systemic Lupus International Collaborating Clinics (SLICC) classification criteria and matched controls.

Exclusion Criteria:

* Co-existing chronic inflammatory or autoimmune diseases.
* Age <18 years
* Malignancy.
* Pregnancy or lactation.
* Chronic liver or renal insufficiency.
* Malignant hematologic diseases.
* Active hepatitis.
* Acute infection within the previous four weeks

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Group 1:patients aged 18 year and older both males and females diagnosed with systemic lupus erythematosus fulfilling the systemic lupus international collaborating clincs (SLICC) admitted to Physical Medicine, Rheumatology and Rehabilitation Department .
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
assess the utility of the albumin-to-globulin ratio (AGR) as reliable, non-invasive biomarker for predicting disease activity in patients with systemic lupus erythematosus (SLE). | From 6 month to one year

CONTACTS AND LOCATIONS:
Overall Officials: Esam M Abualfadl, Professor, Study Chair — Sohag University; Rabab H Ali, MD, Study Director — Sohag University
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Idborg H, Eketjall S, Pettersson S, Gustafsson JT, Zickert A, Kvarnstrom M, Oke V, Jakobsson PJ, Gunnarsson I, Svenungsson E. TNF-alpha and plasma albumin as biomarkers of disease activity in systemic lupus erythematosus. Lupus Sci Med. 2018 Jun 4;5(1):e000260. doi: 10.1136/lupus-2018-000260. eCollection 2018. PMID 29955370
- [Background] Guo X, Shao J, Zhai B, Zou Q, Yan J, Gu H, Wang G. Relationship and prognostic significance between preoperative serum albumin to globulin ratio and CT features of non-small cell lung cancer. Eur J Radiol. 2020 Jul;128:109039. doi: 10.1016/j.ejrad.2020.109039. Epub 2020 May 4. PMID 32417713
- [Background] Barber MRW, Drenkard C, Falasinnu T, Hoi A, Mak A, Kow NY, Svenungsson E, Peterson J, Clarke AE, Ramsey-Goldman R. Global epidemiology of systemic lupus erythematosus. Nat Rev Rheumatol. 2021 Sep;17(9):515-532. doi: 10.1038/s41584-021-00668-1. Epub 2021 Aug 3. PMID 34345022
- [Background] Aringer M, Costenbader K, Daikh D, Brinks R, Mosca M, Ramsey-Goldman R, Smolen JS, Wofsy D, Boumpas DT, Kamen DL, Jayne D, Cervera R, Costedoat-Chalumeau N, Diamond B, Gladman DD, Hahn B, Hiepe F, Jacobsen S, Khanna D, Lerstrom K, Massarotti E, McCune J, Ruiz-Irastorza G, Sanchez-Guerrero J, Schneider M, Urowitz M, Bertsias G, Hoyer BF, Leuchten N, Tani C, Tedeschi SK, Touma Z, Schmajuk G, Anic B, Assan F, Chan TM, Clarke AE, Crow MK, Czirjak L, Doria A, Graninger W, Halda-Kiss B, Hasni S, Izmirly PM, Jung M, Kumanovics G, Mariette X, Padjen I, Pego-Reigosa JM, Romero-Diaz J, Rua-Figueroa Fernandez I, Seror R, Stummvoll GH, Tanaka Y, Tektonidou MG, Vasconcelos C, Vital EM, Wallace DJ, Yavuz S, Meroni PL, Fritzler MJ, Naden R, Dorner T, Johnson SR. 2019 European League Against Rheumatism/American College of Rheumatology classification criteria for systemic lupus erythematosus. Ann Rheum Dis. 2019 Sep;78(9):1151-1159. doi: 10.1136/annrheumdis-2018-214819. Epub 2019 Aug 5. PMID 31383717